CLINICAL TRIAL: NCT04073667
Title: Investigation of the Effects of Exercise Program Applied on Postoperative Period in Patients With Chiari Type 1 Malformation
Brief Title: Investigation of the Effects of Exercise Program in Patients With Chiari Type 1 Malformation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ceyhun Turkmen, Research Assisstant, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KA-19064
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Arnold Chiari Malformation
Keywords: balance; proprioception; exercise; cervical region; chiari malformation; rehabilitation
MeSH Terms: conditions — Arnold-Chiari Malformation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Rehabilitation Group (Experimental): The first six weeks (1st-6th) will be followed as an exercise group and the second six weeks (7th-12th) will be followed as a control group without any intervention.
  Interventions: Behavioral: Exercise
- Late Rehabilitation Group (Experimental): The first six weeks (1st-6th) will be followed as a control group without any intervention and the second six weeks (7th-12th) will be followed by exercise.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Specific Exercises:
  a. Exercises for cervical flexors: Objectives are summarized below:
  * To increase the endurance and strength of cervical flexors. b. Exercises for cervical extensors:
  * Training of craniocervical extensors and rotators with the cervical spine in the neutral position, c. Axiocapular muscles;
  * Teaching the correct scapular position, D. Postural correction exercises;
  * Teaching the neutral spine position from the first treatment session, 2) Sensorimotor Exercises:
    a. Joint position sense:
  * Participants are trained to point their heads in different directions with the help of an illuminated band that is attached to the head with the eyes open at the beginning.
    b. The sense of cervical movement, c. Oculomotor control exercises, 3) Balance and coordination exercises;
    a. Balance training starts with static balance exercises and continues with dynamic balance exercises and walking exercises with different difficulty.

SUMMARY:
This study will be conducted in Hacettepe University Faculty of Medicine Neurosurgery Department and Hacettepe University Faculty of Physical Therapy and Rehabilitation.

The study was designed as a randomized controlled trial. At the beginning of the study, demographic data and characteristics of the cases will be recorded. Patients will be evaluated in three different periods throughout the study. The first assessments will be performed on the first day after the patient's condition is appropriate after the surgical procedure for Type 1 CM. Following this evaluation, all patients will be divided into two groups using. a simple randomization method. The first group will be exercised for 6 weeks while the second group will not be intervened during this period and will be followed as a control group. Immediately after the exercise program administered to the first group after 6 weeks, both groups will undergo second assessments. After these assessment measures, the same exercise program in the first group will be applied to the second group only this time for 6 weeks. In the meantime, the first group will stop their exercise programs. After the 6-week exercise program of the second group has ended, both groups will be given the third assessment, the final assessment.

At the beginning of the study, demographic data, characteristics and disease information will be recorded.

The evaluations to be made are summarized below:

* Visual Analogue Scale, pain threshold and pain tolerance tests, Neck Disability Index, for the determination of pain level in the neck region and throughout the body
* Cervical range of motion (Performance Attainment Associates, St. Paul, MN, 55117, United States) (CROM 3) device for the evaluation of the cervical region.
* Berg Balance Scale for evaluation of performance-based balance,
* Timed Rise Walk Test, Sharpened Romberg test and "8" shaped walk test (F8WT) for evaluation of fall risk, static and dynamic balance,
* The International Ataxia Assessment Scale (ICARS) for coordination,
* Grip Ability Test (GAT) for the assessment of fine motor skill in the upper extremity,
* Posture evaluation,
* Eating Assessment Tool (EAT-10) for evaluation of swallowing function
* For daily living activities, Barthel Daily Living Activities Index,
* For the quality of life, the Short Form 36 questionnaire will be used.

DETAILED DESCRIPTION:
This study will be conducted in Hacettepe University Faculty of Medicine Neurosurgery Department and Hacettepe University Faculty of Physical Therapy and Rehabilitation.

The study was designed as a randomized controlled trial. At the beginning of the study, demographic data and characteristics of the cases will be recorded. Patients will be evaluated in three different periods throughout the study. The first assessments will be performed on the first day after the patient's condition is appropriate after the surgical procedure for Type 1 CM. Following this evaluation, all patients will be divided into two groups using. a simple randomization method. The first group will be exercised for 6 weeks while the second group will not be intervened during this period and will be followed as a control group. Immediately after the exercise program administered to the first group after 6 weeks, both groups will undergo second assessments. After these assessment measures, the same exercise program in the first group will be applied to the second group only this time for 6 weeks. In the meantime, the first group will stop their exercise programs. After the 6-week exercise program of the second group has ended, both groups will be given the third assessment, the final assessment.

"The study will be conducted in individuals aged 18-65 years who have been diagnosed with Type 1 CM by the physician and have been decided to undergo surgery for this diagnosis. In our study whose primary outcome parameters were determined as "Neck Disability Index" and "Visual Analogue Scale minimum, the minimum sample width required to reach 95% -99% power was six individuals in total. For various reasons (patient withdrawal, etc.), the rate of withdrawal from the study was predicted to be 25%. Accordingly, the study was decided to be conducted with a total of eight individuals.

Patients with a history of primary neurological disease other than Chiari Type 1 Malformation, severe cognitive impairment (> 24 from Mini-Mental State Assessment), peripheral vestibular problem, and history of orthopedic surgery will not be included in the study.

The data will be evaluated using SPSS for Windows 22.00. Descriptive statistics will be presented as a minimum, average, median, standard deviation, maximum and categorical variables for numerical variables and as percentages. The suitability of the variables to normal distribution will be examined by the Shapiro-Wilk normality test. Whether the groups (Group 1, Group 2) are similar in terms of gender will be examined by the Pearson Chi-Square Test when the prerequisites are met, and Fisher's exact test if not. By the cross-pass research design, the block, period, trial and sequence effects will be analyzed with a mixed effect model.

At the beginning of the study, demographic data, characteristics and disease information will be recorded.

The evaluations to be made are summarized below:

* Visual Analogue Scale, pain threshold and pain tolerance tests, Neck Disability Index, for the determination of pain level in the neck region and throughout the body
* Cervical range of motion (Performance Attainment Associates, St. Paul, MN, 55117, United States) (CROM 3) device for the evaluation of the cervical region.
* Berg Balance Scale for evaluation of performance-based balance,
* Timed Rise Walk Test, Sharpened Romberg test and "8" shaped walk test (F8WT) for evaluation of fall risk, static and dynamic balance,
* The International Ataxia Assessment Scale (ICARS) for coordination,
* Grip Ability Test (GAT) for the assessment of fine motor skill in the upper extremity,
* Posture evaluation,
* Eating Assessment Tool (EAT-10) for evaluation of swallowing function
* For daily living activities, Barthel Daily Living Activities Index,
* For the quality of life, the Short Form 36 questionnaire will be used.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted in individuals aged 18-65 years who have been diagnosed with Type 1 CM by the physician and have been decided to undergo surgery for this diagnosis.

Exclusion Criteria:

* Patients with a history of primary neurological disease other than Chiari Type 1 Malformation, severe cognitive impairment (> 24 from Mini Mental State Assessment), peripheral vestibular problem, and history of orthopedic surgery will not be included in the study. .

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-11-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | VAS was used to assess changes in chronic and experimental pain of individuals at 6th and 12th week of exercise intervention.
  Visual analogue scales (VAS) of sensory intensity and affective magnitude were validated as ratio scale measures for both chronic and experimental pain.
Neck Disability Index | NDI was used to assess changes in functional status of patients with neck pain at 6th and 12th week of exercise intervention.
  The Neck Pain Disability Index (NDI) is a questionnaire that is commonly used in clinical trials to measure the functional status of patients with neck pain. The NDI was originally developed for assessing the functional status of patients with disabling neck pain, particularly whiplash-associated disorders. The NDI consists of 10 items addressing functional activities, such as personal care, lifting, reading, work, driving or cycling, sleeping and recreational activities, and a number of symptoms such as pain intensity, concentration, and headache.For each item, answering options range from 0 = no disability to 5 = total disability, resulting in a total range of scores from 0 to 50 points.

SECONDARY OUTCOMES:
Berg Balance Scale | BBS was used to assess changes in functional balance performance at 6th and 12th week of exercise intervention.
  The Berg balance scale (BBS) assesses functional balance performance based on 14 items common to daily life. The maximum score that can be reached is 56 and each item possesses an ordinal scale of five alternatives ranging from 0 to 4 points.
Sharpened Romberg Test | Sharpened Romberg Test was used to assess changes in functional balance performance at 6th and 12th week of exercise intervention.
  The subjects were instructed to stand barefoot with the dominant foot just in front of the other (tandem stand, i.e., heel to toe), arms folded across the chest, with eyes open in the first trial, and with eyes closed in a second trial. The score was the number of seconds the subject maintained the test position. Timing started when the subject assumed the proper position and indicated she was ready. Timing stopped if the subject moved either foot from the proper position, opened her eyes in the eyes closed trial, or reached the 60 second time limit.
Short Form 36 | Short Form 36 was used to assess changes in quality of life at 6th and 12th week of exercise intervention.
  The SF36 is a short questionnaire with 36 items which measure eight multi-item variables: physical functioning (10 items), social functioning (two items), role limitations due to physical problems (four items), role limitations due to emotional problems (three items), mental health (five items), energy and vitality (four items), pain (two items), and general perception of health (five items).
Barthel Daily Living Activity Index | Short Form 36 was used to assess changes in daily living activities at 6th and 12th week of exercise intervention.
  Barthel Index of Activities of Daily Living. The Barthel Index (BI) is one of the most widely used rating scales for the measurement of activity limitations in patients with neuromuscular and musculoskeletal conditions in an inpatient rehabilitation setting.

CONTACTS AND LOCATIONS:
Locations (1):
- Ceyhun Türkmen, Ankara, Turkey (Türkiye)